CLINICAL TRIAL: NCT05565989
Title: Alcohol Consumption, Intention Implementation and Mindfulness Meditation (ADUC-Volet 3 " Prevention ")
Acronym: ALCOMEDIIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22-0099
Record Dates: First submitted 2022-09-30; First posted 2022-10-04 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2023-09

CONDITIONS: Binge Drinking; Alcohol Drinking
Keywords: mindfulness; intention implementation; motivationnal interview
MeSH Terms: conditions — Binge Drinking; Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: 1 control condition implying a Motivational Interview (MI)
  1 experimental condition implying a Motivational Interview (MI) + Mindfulness-Based Meditation practices (MBM) + Intention Implementation (II)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (MI) (Active Comparator): Motivational Interview
  Interventions: Behavioral: MI
- experimental (MI/MBM/II) (Experimental): Motivational Interview + mindfulness-bases meditation practice + intention implementation
  Interventions: Behavioral: MBM and II; Behavioral: MI

INTERVENTIONS:
Behavioral: MBM and II — An initiation to MBM practice (including 4 exercices) and 2 intention implementation exercices are proposed to participants
  Arms: experimental (MI/MBM/II)
Behavioral: MI — A motivational Interview will be conducted with participant.

SUMMARY:
The emergence of new problematic alcohol consumption practices among young people requires new dynamics in prevention strategies. In this context, the ADUC project (Alcohol and Drugs at the University of Caen) aims to develop a better understanding of alcohol consumption, and in particular the practice of binge drinking (BD), in order to develop relevant and adapted prevention tools. The ALCOMEDIIT study (IRESP funding; Agreement 20II31-00 - ADUC part 3) is a randomized controlled trial that focuses on the specific determinant of impulsivity. The main objective of this experiment in social psychology is to validate a program for the prevention of BD practices based on motivational interviewing (MI) associated with intention implementation (II) and mindfulness meditation (MBM) in a student environment.

DETAILED DESCRIPTION:
Context. The emergence of new problematic alcohol consumption practices among young people requires new dynamics in prevention strategies. In this context, the ADUC project (Alcohol and Drugs at the University of Caen) aims to develop a better understanding of alcohol consumption, and in particular the practice of binge drinking (BD), in order to develop relevant and adapted prevention tools. The first step, logistically supported by the University of Caen, consisted in identifying the levels of alcohol consumption of students, the prevalence of binge drinking, and their determinants. Based on more than 7000 participants interviewed, it essentially demonstrated 1) an alarming 22% prevalence of BD among students and 2) four main psychological determinants, namely impulsivity (i.e., the tendency of individuals to act prematurely without fully weighing the consequences of their action), subjective norm (i.e., perception of what is done and/or approved by peers), drinker identity (i.e., how the individual defines him/herself as a drinker), and motivations to drink (social, compliance, enhancement, or coping motivations).

Objective. The ALCOMEDIIT study (IRESP funding; Agreement 20II31-00 - ADUC part 3) is a randomized controlled trial that focuses on the specific determinant of impulsivity. The main objective of this experiment in social psychology is to validate a program for the prevention of BD practices based on motivational interviewing (MI) associated with intention implementation (II) and mindfulness meditation (MBM) in a student environment.

Materials and Methods. This study will include 120 healthy subjects who will be students at the University of Caen Normandy. They will be people who consume alcohol, having a BD score > 1 in the month preceding the inclusion but not presenting any specific disorder. The trial will be proposed to them by e-mail and the people who meet the inclusion criteria will join either a control group which will benefit from a MI, or an experimental group which will also benefit from a MI but which will be associated with an initiation to MBM with II (initial visit T0). In order to measure the effectiveness of the prevention device in terms of reducing the use of BD, a follow-up at 1 month (T1) as well as a follow-up at 6 months (T6; exploratory) will be proposed to all participants. The total duration of this research protocol is one year.

Hypothesis tested. The aim of this work is to evaluate the interest of associating mindfulness meditation practices, practices implemented to optimize their use, with a motivational interview in a prevention program aiming at reducing alcohol use and the practice of BD in the student population.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 30 years old,
* of French mother language,
* of both sexes,
* binge drinking score > 1,
* having signed an informed consent.

Exclusion Criteria:

* Pregnant or breastfeeding students,
* students who declare a history of neurological, neurosurgical, psychiatric, endocrine or infectious diseases.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
binge drinking score | 1 month
  The BD score (Townshend & Duka, 2005) is calculated on the basis of 3 distinct elements (Q1: "number of average standard drinks per hour (containing about 10g of pure alcohol in France)"; Q2: "number of drunken episodes in the last month" and Q3; "percentage of drunken episodes among the occasions of drinking"). The score results from the following weighting: (4 x Q1) + Q2*6 + (0.2 x Q3). This score considers both the quantity and frequency of drinking, thus integrating the dimension of repeated alcohol withdrawal.

SECONDARY OUTCOMES:
craving | 1 month
  1 item measuring craving
craving | 6 months
  1 item measuring craving
impulsivity | 1 month
  UPPS Scores
impulsivity | 6 months
  UPPS Scores
Readiness to Change Alcohol consumption | 1 month
  This self-assessment based on the transtheoretical model of behaviour change (Prochaska & DiClemente, 1982, DiClemente & Prochaska, 1982) is recognized for its reliability and validity. The RTC-Alcohol has three different scales that correspond to an assessment of the three main stages of behaviour change: the pre-contemplation, contemplation and action stages. Based on the person's score on each of these scales, the experimenter determines which stage of behavior change the person is in.
Readiness to Change Alcohol consumption | 6 months
  This self-assessment based on the transtheoretical model of behaviour change (Prochaska & DiClemente, 1982, DiClemente & Prochaska, 1982) is recognized for its reliability and validity. The RTC-Alcohol has three different scales that correspond to an assessment of the three main stages of behaviour change: the pre-contemplation, contemplation and action stages. Based on the person's score on each of these scales, the experimenter determines which stage of behavior change the person is in.
alcohol use | 6 month
  number of alcoholic drinks
binge drinking score | 6 month
  The BD score (Townshend & Duka, 2005) is calculated on the basis of 3 distinct elements (Q1: "number of average standard drinks per hour (containing about 10g of pure alcohol in France)"; Q2: "number of drunken episodes in the last 6 months" and Q3; "percentage of drunken episodes among the occasions of drinking"). The score results from the following weighting: (4 x Q1) + Q2 + (0.2 x Q3). This score considers both the quantity and frequency of drinking, thus integrating the dimension of repeated alcohol withdrawal.
Alcohol use | 1 month
  Number of alcoholic drinks

CONTACTS AND LOCATIONS:
Overall Officials: Jessica MANGE, PhD, Principal Investigator — University of Caen Normandy
Locations (1):
- University of Caen Normandy, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: No
Study protocol and statistical analysis plan will be shared.

REFERENCES:
- [Derived] Mange J, Mauny N, Montcharmont C, Legrand E, Lemercier-Dugarin M, Mortier A, Duvivier M, Leveneur J, Lacherez C, Cabe N, Le Berre AP. A prevention program for binge drinking among students based on mindfulness and implementation intention (ALCOMEDIIT): a randomized controlled trial. Trials. 2024 Jan 2;25(1):1. doi: 10.1186/s13063-023-07887-9. PMID 38169391